CLINICAL TRIAL: NCT04494308
Title: Pilot Study for Evaluation of Eosinophils Phenotype and Activation Status in COPD Patients
Brief Title: Evaluation of Eosinophil Phenotype in COPD Patients
Acronym: V-FEO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS San Raffaele Roma (Other)
Responsible Party: Sponsor
Other Study IDs: RP 06/18
Record Dates: First submitted 2020-07-28; First posted 2020-07-31 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2023-06

CONDITIONS: COPD; COPD Exacerbation
Keywords: eosinophils; immunophenotype; inflammation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exacerbated: COPD patients admitted to the hospital for an exacerbation occurred within the past 10 days.
  Interventions: Other: biomarker identification
- stable: COPD stable patients with no exacerbations in the past 3 months
  Interventions: Other: biomarker identification

INTERVENTIONS:
Other: biomarker identification — flow cytometric analysis of eosinophils membrane molecules

SUMMARY:
This is a pilot non pharmacological observational study. Aim of the study is to analyze the immunophenotype of circulating eosinophils in chronic obstructive pulmonary disease (COPD) patients, and to correlate results with clinical status of patients (stable versus exacerbated patients, response to therapy). In about 30% of COPD patients there is an increase in the number of circulating eosinophils, which associates with an increased risk for exacerbation. However, no data is available on the role of eosinophils in this disease, on their activation status and their response to chemotactic factors. By multicolor flow cytometry the investigators will analyze membrane molecules and intracellular cytokines associated to chemotaxis, degranulation and inflammation. The study will enroll 30 patients (15 stable and 15 with exacerbation). Results will be analyzed taking into account clinical status,disease progression and response to treatment.

DETAILED DESCRIPTION:
In about 30% of COPD patients there is an increased number of circulating eosinophils. On their membrane, eosinophils express several molecules, also related to their physiology, namely major histocompatibility complex (MHC) class II, needed for antigen presentation; CCR3, receptor for a variety of chemokines, including eotaxin (CCL11), eotaxin-3 (CCL26), monocyte chemotactict protein (MCP)-3 (CCL7), MCP-4 (CCL13), and RANTES (CCL5); cluster of differentiation (CD)125, which binds IL-5 and stimulates eosinophils proliferation; CD63, a marker that is upregulated after eosinophils degranulation; and CD294 (CRTH2) which is the prostaglandin D2 receptor, and is associated to allergy and inflammation . The hypothesis for the present trial is that different clinical phenotypes of COPD patients could be associated to different activation statuses of eosinophils, that can be evaluated analyzing by flow cytometry the membrane expression of the above mentioned molecules. In particular, the investigators hypothesize that membrane molecules may be modulated in different stages of the diseases, and may change after medical and rehabilitative therapies.

The investigators will analyze phenotype of eosinophils from blood samples of patients with COPD, admitted to the hospital after an episode of exacerbation, or for routine controls. In this way, the association between a particular pattern of molecules expressed on eosinophils membrane and the severity of COPD will be defined. Moreover, for hospitalized patients, eosinophils phenotype also on discharge day will be analyzed. In this way the effect of therapies on eosinophils activation will be assessed. Clinical status of patients will be assessed by standard tests such as St George Respiratory Questionnaire (SGRQ), BODE index, COPD Assessment Test (CAT), Six min. Walking Test (6'WT), Pulmonary Function Tests (PFT).

Eosinophils phenotype and in vitro cytokines production will be analyzed by multicolor flow cytometry. To minimize the effect of manipulation, staining of membrane molecules will be performed on whole blood samples, followed by lysis of erythrocytes. The following molecules will be analyzed: CD45, CD16, CD15, CD63, CCR3, CD125, CD294, Siglec-8. After in vitro stimulation with lipopolysaccharide (LPS) or CCL11, the production of interleukine (IL)-4, TGFbeta and IL-2 will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* percentage of eosinophils >0%
* episode of exacerbation in the previous 10 days (for exacerbated cohort)
* no exacerbation in the previous 3 months (for stable cohort)

Exclusion Criteria:

* percentage of eosinophils =0%
* history of allergic diseases
* patients that are currently enrolled in other clinical trials involving new drugs or treatments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 COPD patients, of which 15 will be COPD patients admitted to the Pulmonary Rehabilitation Unit of IRCCS San Raffaele Pisana hospital for an exacerbation occurred within the past 10 days (exacerbated cohort); the other 15 will be stable patients, (no exacerbations in the past 3 months- stable cohort), affering to the hospital as outpatients for routine controls
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Association of eosinophils phenotype with clinical status in COPD patients | one year
  We expect to identify different patterns of expression of molecules on eosinophils membrane that are associated with different clinical phenotypes of COPD patients. We will also associate eosinophils phenotype to the response to medical and rehabilitation therapy. The definition of these patterns will provide a diagnostic tool to rapidly identify patients that will benefit from a specific therapy

CONTACTS AND LOCATIONS:
Overall Officials: Laura Vitiello, PhD, Principal Investigator — IRCCS San Raffaele Pisana, Roma
Locations (1):
- IRCCS San Raffaele Pisana, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No